CLINICAL TRIAL: NCT06713499
Title: A Phase Ib/II Study to Investigate the Safety、PK and PD of SHR-1819 in Children and Adolescents With Moderate-to-severe Atopic Dermatitis
Brief Title: A Phase Ib/II Study to Investigate the Safety of SHR-1819 in Children and Adolescents With Moderate-to-severe Atopic Dermatitis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1819-204
Record Dates: First submitted 2024-11-24; First posted 2024-12-03 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Children and Adolescents With Moderate-to-severe Atopic Dermatitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1819 injection (Experimental): Dose 1, dose 2 and dose 3.
  Interventions: Drug: SHR-1819 injection

INTERVENTIONS:
Drug: SHR-1819 injection — SHR-1819 injection.

SUMMARY:
This trial was designed to evaluate the safety of SHR-1819 in children and adolescents with moderate-to-severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects and their parents or legal guardians have voluntarily signed the informed consent form prior to the start of any procedures related to the study, are able to communicate smoothly with the investigator, understand and are willing to strictly comply with the requirements of this clinical study protocol to complete the study;
2. At the time of signing the informed consent, the subjects were ≥ 6 years old and < 18 years old, male or female;
3. Have atopic dermatitis at screening.

Exclusion Criteria:

1. Before enrollment, the subjects weighed < 15kg;
2. Females who are pregnant or lactating and have a positive pregnancy test result;
3. Have other active skin disease or skin complications due to other conditions that may affect the evaluation of AD;
4. Have serious concomitant diseases and other conditions that the investigator considers inappropriate to participate in this trial;
5. Treated with biologics targeting IL-4Rα , or participated in previous clinical studies of biologics targeting IL-4Rα, including SHR-1819 injection;
6. Has malignancy or has a history of malignancy;
7. Hypersensitivity to the study drug or any ingredient in the study drug.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Up to 14 weeks.
Heart rate | Up to 14 weeks.
PR interval | Up to 14 weeks.
QT interval | Up to 14 weeks.
QRS duration | Up to 14 weeks.

SECONDARY OUTCOMES:
The concentration of SHR-1819 in serum | From the beginning of administration to the 14th week.
Changes in the level of TARC/CCL17 in the serum | From the beginning of administration to the 14th week.
  Changes in the level of biomarkers in serum.
Evaluate the incidence and timing of ADA positivity for SHR-1819 | From the beginning of administration to the 14th week.
  Changes in the level of immunogenicity in the body.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided